CLINICAL TRIAL: NCT02663349
Title: Skills Training to Enhance Vocational Outcomes in Veterans With Serious Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Minnesota Veterans Medical Research and Education Foundation (Other)
Responsible Party: Principal Investigator, Tasha Nienow, Principal Investigator, Minneapolis Veterans Affairs Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4612-A
Record Dates: First submitted 2016-01-19; First posted 2016-01-26 (Estimated); Results first posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2022-06

CONDITIONS: Schizophrenia; Bipolar Disorder; Psychotic Disorders
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Supported SCIT (Experimental): Social Cognition and Interaction Training is a manualized intervention that focuses on emotion recognition training, perspective taking, and strategies to avoid jumping to conclusions. One 2-hour group session will be offered once a week for 12 weeks. In addition, 30 minutes of individual training will be provided weekly by an instructor.
  Interventions: Behavioral: Social Cognition and Intervention Training

INTERVENTIONS:
Behavioral: Social Cognition and Intervention Training — A manualized group therapy that teaches social cognitive skills.

SUMMARY:
Maintenance of employment is dependent upon being able to successfully integrate into one's work setting. This can present a significant challenge to individuals with serious mental illness, as they typically exhibit impairment in their ability to accurately perceive and understand social exchanges. Presently the most established intervention is Social Cognition and Interaction Training (SCIT), a 12-week group intervention in which participants learn strategies to enhance emotion recognition and to assess the accuracy of their interpretation of social interactions. To enhance transfer of training gains to functional outcomes, participants will be paired with a social mentor to facilitate completion of homework and to ensure that skills are practiced outside of treatment (supported SCIT). The study will examine the impact of supported SCIT on social and work role functioning.

The specific aims are:

1. To assess the feasibility of providing supported SCIT to individuals with serious mental illness who are engaged in compensated work activity.
2. To assess the impact of supported SCIT on social cognitive skills as well as work and social performance.
3. To assess durability of intervention-induced change 3 months after the end of intervention.

A single blind study will be conducted in which participants between 18-70 with serious mental illness (schizophrenia, schizoaffective disorder, and bipolar disorder) are assigned to 12 weeks of supported SCIT. Intervention will consist of one 2-hour small group training sessions and 30 minutes of individualized supported practice of skills with a treatment facilitator weekly. Feasibility will be assessed with attendance at group and individual sessions. Baseline, post-intervention (3-month), and follow-up (6-month) assessments will measure social cognitive abilities and functional outcomes. Potentially confounding variables such as symptom severity and outside treatment hours will also be assessed. It is hypothesized that supported SCIT will be completed by at least 75% of veterans. The intervention is predicted to improve social cognitive skills and social and work performance. Training gains are expected to be sustained 3 months after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Schizophrenia, Schizoaffective Disorder, or Bipolar Disorder
* Veteran
* Engaged in compensated work activity, volunteer work, school
* Age 18 to 70

Exclusion Criteria:

* Currently meet criteria for substance abuse or have met criteria for substance dependence in that previous 6 months
* Have an estimated premorbid IQ below 70,
* Have a history of a clinically significant head injury or neurological disease
* Do not speak English well enough to comprehend testing procedures
* Do not demonstrate adequate understanding of study procedures to give informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tasha M Nienow, PhD, Principal Investigator — Minneapolis Veterans Affairs Medical Center
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment was conducted at the Minneapolis VA Health Care System (VAHCS) between January 2016 and October 2017. Letters describing the study were sent to veterans enrolled at the Minneapolis VAHCS who had a diagnosis of a psychotic or mood disorder. Veterans were given 2 weeks to respond to the letter. When veterans did not respond, research staff contacted them by phone to ask about their interest in the study.
Pre-assignment Details: Participants were not excluded after enrollment in the study. Several enrolled participants chose not to participate when they were informed of their eligibility, citing being too busy, changes in schedule, or new plans to move out of the area.
Groups:
- Supported SCIT: Social Cognition and Interaction Training is a manualized intervention that focuses on emotion recognition training, perspective taking, and strategies to avoid jumping to conclusions. One 2-hour group session was offered once a week for 12 weeks. In addition, 30 minutes of individual training was provided weekly by an instructor.
  Social Cognition and Intervention Training: A manualized group therapy that teaches social cognitive skills.
Period: Overall Study
Arm/Group | Supported SCIT
Started | 22
Attended First Treatment Session | 18
Completed Intervention | 16
Completed Follow-up Assessment 3 Months Post-intervention | 16
Completed | 16
Not Completed | 6
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Population: Analysis was done only with participants who completed the study. Baseline data is for the 16 participants who completed the study.
Arm/Group | Supported SCIT
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.62 (10.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16
Years of Education [Mean (Standard Deviation); unit: years] | 15.13 (1.59)
Wechsler Test of Adult Reading Estimated Full Scale IQ [Mean (Standard Deviation); unit: units on a scale] — Wechsler Test of Adult Reading (WTAR) Estimated Premorbid Intellectual Function
  This is a measure of intellectual function prior to the onset of illness or disease. Score ranges from 64-124. Higher scores mean better intellectual functioning. A score of 100 is considered average.
  units on a scale | 105.94 (6.51)
Brief Psychiatric Rating Scale Total score [Mean (Standard Deviation); unit: units on a scale] — This is 24 item measure of psychiatric symptom severity. Each item can be rated from 1 (not present) to 7 (extremely severe). Total score scale range is 24-168 with a higher score indicating presence of more severe psychiatric symptoms.
  units on a scale | 36.00 (7.84)
Length of Illness in years [Mean (Standard Deviation); unit: years] | 26.38 (10.99)

OUTCOME MEASURES:

1. Primary Outcome: Bell-Lysaker Emotion Recognition Task Total Score
Description: This task measures emotion recognition ability. Total score ranges from 0-21. A higher score indicates better performance.
Time Frame: Total score at Baseline and 3 months
Population: One participant produced invalid results on this measure and their data was removed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supported SCIT
Number analyzed (Participants) | 15
score on a scale
  Baseline | 14.8 (3.10)
  3 month assessment | 16.00 (2.42)
Statistical Analysis 1: Comparison: Supported SCIT; Within sample analysis of change between baseline and 3 month assessment; Test type: Superiority; p = .08, t-test, 2 sided; df = 14

2. Primary Outcome: Bell-Lysaker Emotion Recognition Task Total Score
Description: as for outcome 1
Time Frame: Total score at Baseline and at 6 months
Population: One participant produced invalid results on this measure and their data was removed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supported SCIT
Number analyzed (Participants) | 15
score on a scale
  Baseline | 14.8 (3.10)
  6 month assessment | 15.13 (3.27)
Statistical Analysis 1: Comparison: Supported SCIT; Within sample change between baseline and 6 month assessment; Test type: Superiority; p = .69, t-test, 2 sided

3. Primary Outcome: Facial Emotion Identification Test Total Score
Description: This is a measure of emotion recognition. Total score ranges from 0-19. A higher score indicates better emotion recognition ability.
Time Frame: Total score at Baseline and at 3 months
Population: completer analysis, Scores for one participant were removed for this measure due to invalid performance.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supported SCIT
Number analyzed (Participants) | 15
score on a scale
  Baseline Assessment | 12.20 (3.26)
  3-month Assessment | 13.8 (2.60)
Statistical Analysis 1: Comparison: Supported SCIT; Within sample change assessed between baseline and 3-month assessment; Test type: Superiority; p = .02, t-test, 2 sided; df=14

4. Primary Outcome: Facial Emotion Identification Test Total Score
Description: This is a measure of emotion recognition ability. Scores range from 0-19. A higher score indicates better performance.
Time Frame: Total score at Baseline and at 6 months
Population: completer analysis, Scores from one participant were removed from this analysis due to invalid performance.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supported SCIT
Number analyzed (Participants) | 15
score on a scale
  Baseline Assessment | 12.20 (3.26)
  6 Month Assessment | 12.4 (3.07)
Statistical Analysis 1: Comparison: Supported SCIT; Change between baseline and 6 month assessment; Test type: Superiority; p = .34, t-test, 2 sided; df = 14

5. Primary Outcome: Ambiguous Intentions and Hostility Scale - Hostility and Aggression Total Scores
Description: The Hostility Total score is a measure of attributional bias and reflects the amount of hostility that is perceived in the actions of others when a situation is ambiguous. Score ranges from 1 (Not at all Hostile, An accident) to 5 (Very Hostile, the other person intended to hurt me) A higher score indicates greater hostility is perceived.
  The Aggression Total score is a measure of how aggressively a participant reports that they would respond to an ambiguous situation in which they are mistreated. Score ranges from 1 (Not at all Aggressive, participant says he would do nothing) to 5 (Very Aggressive, participant would retaliate physically). A 1 is a passive response, a 3 is an assertive response, and a 5 is a very aggressive response.
Time Frame: Total score at Baseline and at 3 months
Population: completer analysis of AIHQ Hostility and Aggression scale Total scores
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supported SCIT
Number analyzed (Participants) | 16
score on a scale
  Baseline AIHQ Hostility scale | 2.20 (.70)
  3-Month Assessment AIHQ Hostility scale | 2.09 (.58)
  Baseline AIHQ Aggression scale | 1.61 (.29)
  3-Month Assessment AIHQ Aggression scale | 1.84 (.45)
Statistical Analysis 1: Comparison: Supported SCIT; completer analysis of change between baseline and 3-month assessment on the AIHQ Hostility scale; Test type: Superiority; p > .05, t-test, 2 sided
Statistical Analysis 2: Comparison: Supported SCIT; Completer analysis to examine within group change between baseline and 3-month assessment on the AIHQ Aggression scale; Test type: Superiority; p = .04, t-test, 2 sided

6. Primary Outcome: Ambiguous Intentions and Hostility Scale -Hostility and Aggression Scale Total Scores
Description: as for outcome 5
Time Frame: Total score at Baseline and at 6 months
Population: completer analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supported SCIT
Number analyzed (Participants) | 16
score on a scale
  Baseline Assessment AIHQ Hostility scale | 2.20 (.70)
  6-Month Assessment AIHQ Hostility scale | 2.13 (.62)
  Baseline Assessment AIHQ Aggression scale | 1.61 (.29)
  6 Month Assessment Assessment AIHQ Aggression scale | 1.79 (.58)
Statistical Analysis 1: Comparison: Supported SCIT; completer analysis of within group change on the AIHQ Hostility scale between baseline and the 6-month assessment; Test type: Superiority; p > .05, t-test, 2 sided
Statistical Analysis 2: Comparison: Supported SCIT; completer analysis of within group change on the AIHQ Aggression scale between baseline and the 6 month assessment; Test type: Superiority; p > .05, t-test, 2 sided

7. Primary Outcome: The Awareness of Social Inference Test Total Score for Part 3
Description: The Awareness of Social Inference Test (TASIT) total score for Part 3 is a measure of a person's ability to perceive social inferences involved in the telling of lies and the use of sarcasm. The total score ranges from 0 to 64. A higher score indicates better social inference performance.
Time Frame: Total score at Baseline and at 3 months
Population: completer analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supported SCIT
Number analyzed (Participants) | 16
score on a scale
  Baseline Assessment | 49.25 (5.69)
  3 Month Assessment | 47.88 (7.62)
Statistical Analysis 1: Comparison: Supported SCIT; Change within group between baseline and 3 month assessment on the TASIT total score for part 3; Test type: Superiority; p > .05, t-test, 2 sided; df = 15

8. Primary Outcome: The Awareness of Social Inference Task Total Score on Part 3
Description: as for outcome 7
Time Frame: Total score at Baseline and at 6 months
Population: completer analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supported SCIT
Number analyzed (Participants) | 16
score on a scale
  Baseline Assessment | 49.25 (5.69)
  6 Month Assessment | 48.69 (7.45)
Statistical Analysis 1: Comparison: Supported SCIT; within group change on the TASIT total score for Part 3 between baseline and the 6 month assessment; Test type: Superiority; p > .05, t-test, 2 sided; df = 15

9. Secondary Outcome: Social Skill Performance Assessment Total Score
Description: The Total score is a measure of social skill demonstrated in two role plays of everyday social situations. Total score can range from 17-85. A higher score indicates more skillful performance.
Time Frame: Total score at Baseline and at 3 months
Population: Completer analysis. One participant was removed for this measure because they did not cooperate with the role play and produced invalid results.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supported SCIT
Number analyzed (Participants) | 15
score on a scale
  Baseline Assessment | 4.16 (.46)
  3-month assessment | 4.13 (.30)
Statistical Analysis 1: Comparison: Supported SCIT; Within group change on SSPA Total Score between baseline and 3-month assessment; Test type: Superiority; p > .05, t-test, 2 sided; df = 14

10. Secondary Outcome: Social Skill Performance Assessment Total Score
Description: as for outcome 9
Time Frame: Total score at Baseline and at 6 months
Population: Completer analysis. One participant was removed from this analysis because he did not cooperate with the role play and produced invalid results
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supported SCIT
Number analyzed (Participants) | 15
score on a scale
  Baseline Assessment | 4.16 (.46)
  6 Month Assessment | 4.20 (.31)
Statistical Analysis 1: Comparison: Supported SCIT; Within group change on the SSPA total score between baseline and 6 month assessment; Test type: Superiority; p > .05, t-test, 2 sided; df = 14

11. Secondary Outcome: First Episode Social Functioning Scale Performance Total Score on Scales 1-7
Description: Self-report measures of social and community functioning in the past 3 month in the following domains: independent living skills, interacting with people, social activities, intimacy, friendships, family relationships and work. Score reflects participant's report of the frequency with which they engaged in behavior. Total score is a sum of items that range from 1 to 4. The Total score range is 28-112, with a higher score indicating better social functioning in the community.
Time Frame: Total score at Baseline and at 3 months
Population: Completer analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supported SCIT
Number analyzed (Participants) | 16
score on a scale
  Baseline Assessment | 78.88 (9.40)
  3-Month Assessment | 78.69 (7.16)
Statistical Analysis 1: Comparison: Supported SCIT; Within group change on the First Episode Social Functioning Scale Performance Total score on scales 1-7 between baseline and 3-month follow-up; Test type: Superiority; p > .05, t-test, 2 sided; df = 15

12. Secondary Outcome: First Episode Social Functioning Scale Performance Total Score on Scales 1-7
Description: as for outcome 11
Time Frame: Total Score at Baseline and at 6 months
Population: Completer analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supported SCIT
Number analyzed (Participants) | 16
score on a scale
  Baseline Assessment | 78.88 (9.40)
  6-Month Assessment | 77.19 (11.88)
Statistical Analysis 1: Comparison: Supported SCIT; Within group change between baseline and 6-month assessment on the First Episode Social Functioning Scale Performance total score on scales 1-7; Test type: Superiority; p > .05, t-test, 2 sided; df = 15

13. Secondary Outcome: Mentoring and Communication Support Scale Subscale Total Scores
Description: The Mentoring and Communication Support Scale is a self-report measure of perceived relationship quality with colleagues and supervisors at work. The scale has four subscales: Collegial Support, Task Support, Career Mentoring, and Coaching. Collegial Support and Task Support scales indicate the amount of support perceived from co-workers, emotionally and in terms of conveying knowledge about how to do the job. The scales range from 4-20 with a higher score indicating a greater level of perceived support. Career Mentoring and Coaching scales measure support perceived from supervisor in terms of advice as well as instruction on how to do one's job. The Career Mentoring scale ranges from 4-20, with a higher score indicating more support. The Coaching scale ranges from 3-15, with a higher score indicating more support.
Time Frame: Total scores at Baseline and at 3 months
Population: Completer analysis. Two participants could not provide data for this measure, as they worked alone at their jobs.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supported SCIT
Number analyzed (Participants) | 14
score on a scale
  Baseline Assessment MCSS Collegial Support scale | 12.36 (2.62)
  3-Month Assessment MCSS Collegial Support scale | 13.43 (3.06)
  Baseline Assessment MCSS Task Support scale | 14.64 (2.76)
  3-Month Assessment MCSS Task Support scale | 15.36 (2.06)
  Baseline Assessment MCSS Mentor scale | 13.93 (4.09)
  3-Month Assessment MCSS Mentor scale | 13.86 (3.37)
  Baseline Assessment MCSS Coach scale | 8.07 (2.67)
  3-Month Assessment MCSS Coach scale | 8.50 (2.93)
Statistical Analysis 1: Comparison: Supported SCIT; Within group change on the MCSS Collegial Support scale between Baseline and 3-Month assessments; Test type: Superiority; p = .15, t-test, 2 sided; df = 13
Statistical Analysis 2: Comparison: Supported SCIT; Within group change on the MCSS Task Support scale between baseline and 3-month assessments; Test type: Superiority; p = .10, t-test, 2 sided; df = 13
Statistical Analysis 3: Comparison: Supported SCIT; Within group change on the MCSS Mentor scale between baseline and the 3-month assessment; Test type: Superiority; p > .05, t-test, 2 sided; df = 13
Statistical Analysis 4: Comparison: Supported SCIT; Within group change on the MCSS Coach scale between baseline and the 3 month assessment; Test type: Superiority; p > .05, t-test, 2 sided; df = 13

14. Secondary Outcome: Mentoring and Communication Support Scale Subscale Total Scores
Description: as for outcome 13
Time Frame: Total score at Baseline and at 6 month assessments
Population: Completer analysis. Two participants could not provide data on this measure because they worked alone.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supported SCIT
Number analyzed (Participants) | 14
score on a scale
  Baseline Assessment MCSS Collegial Support scale | 12.36 (2.62)
  6-Month Asessment MCSS Collegial Support scale | 14.50 (2.53)
  Baseline Assessment MCSS Task Support scale | 14.64 (2.76)
  6-Month Assessment MCSS Task Support scale | 15.86 (2.21)
  Baseline Assessment MCSS Mentor scale | 13.93 (4.09)
  6-Month Assessment MCSS Mentor scale | 13.07 (4.39)
  Baseline Assessment MCSS Coach scale | 8.07 (2.67)
  6-Month Assessment MCSS Coach scale | 8.29 (2.70)
Statistical Analysis 1: Comparison: Supported SCIT; Within group change on the MCSS Collegial Support scale between baseline and the 6-month assessment; Test type: Superiority; p = .01, t-test, 2 sided; df = 13
Statistical Analysis 2: Comparison: Supported SCIT; Within group change on the MCSS Task Support scale between baseline and 6-month assessment; Test type: Superiority; p = .03, t-test, 2 sided; df = 13
Statistical Analysis 3: Comparison: Supported SCIT; Within group change on the MCSS Mentor scale between baseline and the 6-month assessment; Test type: Superiority; p > .05, t-test, 2 sided; df = 13
Statistical Analysis 4: Comparison: Supported SCIT; Within group change on the MCSS Coach scale between baseline and the 6-month assessment; Test type: Superiority; p > .05, t-test, 2 sided; df = 13

15. Secondary Outcome: Vocational Efficacy in Trauma Survivors Scale Self Disclosure and Workplace Coping Total Scores
Description: The Vocational Efficacy in Trauma Survivors Scale is a self-report measure of perceived social support and efficacy coping with mental health symptoms at work. The scale has two subscales Self Disclosure and Workplace Coping. The Self Disclosure subscale ranges from 4-20, with a higher score indicating greater comfort self disclosing about mental health issues at work. The Workplace Coping subscale ranges from 7-35, with a higher score indicating greater confidence in one's abilities to manage mental health symptoms at work.
Time Frame: Total score at Baseline and at 3 months
Population: Completer analysis. Two participants were not able to provide data on this measure, as they worked alone.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supported SCIT
Number analyzed (Participants) | 14
score on a scale
  Baseline VETSS Self Disclosure scale | 13.14 (3.48)
  3-Month Assessment VETSS Self Disclosure scale | 14.29 (3.25)
  Baseline VETSS Workplace Coping scale | 24.00 (4.82)
  3-Month VETSS Workplace Coping scale | 25.36 (4.14)
Statistical Analysis 1: Comparison: Supported SCIT; Within group change on the VETSS Self Disclosure scale between Baseline and 3-Month Assessment; Test type: Superiority; p = .09, t-test, 2 sided; df = 13
Statistical Analysis 2: Comparison: Supported SCIT; Within group change on the VETSS Workplace Coping scale between Baseline and 3-Month Assessment; Test type: Superiority; p = .12, t-test, 2 sided; df = 13

16. Secondary Outcome: Vocational Efficacy in Trauma Survivors Scale Self Disclosure and Workplace Coping Subscale Total Scores
Description: as for outcome 15
Time Frame: Total score at Baseline and at 6 months
Population: Completer analysis. Two participants were not able to provide data for this measure, as they worked alone.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supported SCIT
Number analyzed (Participants) | 14
score on a scale
  Baseline VETSS Self Disclosure subscale score | 13.14 (3.48)
  6-Month Assessment VETSS Self Disclosure | 24.00 (4.82)
  Baseline VETSS Workplace Coping subscale score | 12.48 (3.61)
  6-Month VETSS Workplace Coping | 24.00 (3.86)
Statistical Analysis 1: Comparison: Supported SCIT; Within group change on VETSS Self Disclosure scale between Baseline and 6 month assessment; Test type: Superiority; p > .05, t-test, 2 sided; df = 13
Statistical Analysis 2: Comparison: Supported SCIT; Within group change on VETSS Workplace Coping scale between baseline and the 6 month assessment; Test type: Superiority; p > .05, t-test, 2 sided; df = 13

17. Other Pre Specified Outcome: Percentage of Participants With Completion of the Training Protocol
Description: Percentage of participants who began the intervention and completed the 3-month training protocol
Time Frame: 3-months
Measure: Count of Participants; unit: Participants
Arm/Group | Supported SCIT
Number analyzed (Participants) | 18
Participants | 16

ADVERSE EVENTS:
Time Frame: For each participant, adverse event data were collected through study completion, an average of 8 months for each participant.
Arm/Group | Supported SCIT
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/49/NCT02663349/Prot_SAP_000.pdf